CLINICAL TRIAL: NCT02530931
Title: Evaluation of Inner Ear and Brain Structures With Contrast-enhanced MRI in Patients With Meniere's Disease
Acronym: PROSPER
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Recruitment problem-covid
Sponsor: University Hospital, Grenoble (Other)
Collaborators: Guerbet (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 38RC15.173
Record Dates: First submitted 2015-08-18; First posted 2015-08-21 (Estimated); Last update posted 2020-11-18 (Actual); Status verified 2020-11

CONDITIONS: Meniere's Disease
MeSH Terms: conditions — Meniere Disease | interventions — Gadolinium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- patients with Meniere's disease (Experimental)
  Interventions: Drug: Gadolinium

INTERVENTIONS:
Drug: Gadolinium — diffusion of gadolinium for a population with Meniere's disease in order to develop an imaging disease screening test

SUMMARY:
* This prospective study aims to better characterize inner ear's perilymphatic structures with Magnetic Resonance Imaging using contrast media and delayed injection in patient's with Meniere's disease.
* MR Perfusion Imaging will be assess in both cochlea as well
* Primary auditory brain pathways will be evaluated through MR diffusion imaging

ELIGIBILITY:
Inclusion Criteria:

* Major subjects of over 40 years (mean age of Meniere's disease 40 to 50 years)
* Informed consent signed
* Medical examination performed prior to participation in research
* Patients with clinical criteria of Meniere's disease according to the classification of the American Association of Otology (ie the combination of a sensorineural hearing loss at low frequencies, recurrent vertigo and tinnitus and / or clogged ear sensation)
* Recipient of a French social security scheme

Exclusion Criteria:

* Patients minors
* Patients on a legal protection regime type guardianship
* Respiratory pathologies, cardiovascular, renal, diabetes
* Claustrophobia
* Contraindications to exposure to a magnetic field
* Contraindications to injecting Dotarem ®

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2016-03-16 (Actual); Primary Completion 2020-09 (Actual); Study Completion 2020-09 (Actual)

PRIMARY OUTCOMES:
Gadolinium enhancement in inner ear structures as measured by MR T1 Weighted-Imaging dynamic measurement | One MR scan (4 hours)

CONTACTS AND LOCATIONS:
Overall Officials: Arnaud ATTYE, PH, Principal Investigator — University Hospital, Grenoble
Locations (1):
- GrenobleUniversityHospital, Grenoble, France